CLINICAL TRIAL: NCT00418119
Title: Phase 4 Study on the Efficacy of Erythropoietin Treatment in Patients With Systolic Left Ventricular Dysfunction, Mild Anemia and Normal Renal Function
Brief Title: Erythropoietin Treatment in Patients With Systolic Left Ventricular Dysfunction, Mild Anemia and Normal Renal Function
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4273
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2006-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Erythropoietin

INTERVENTIONS:
Drug: erythropoietin

SUMMARY:
Erythropoietin Treatment in Patients with systolic left ventricular dysfunction, mild anemia and normal renal function

ELIGIBILITY:
Inclusion Criteria:

* Ischemic heart disease
* Systolic lv dysfunction
* Mild anemia
* Normal renal function
* Stable condition

Exclusion Criteria:

* Pregnancy
* Unstable condition
* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2007-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Tuvia Ben Gal, MD, Principal Investigator — Cardiology Department Rabin medical Center; Ofer Shpilberg, Prof., Study Director — Hematology Department Rabin Medical Center; Daniel Murninkas, MD, Study Director — Cardiology Department Rabin Medical Center
Locations (1):
- Cardiology Department, Rabin Medical Center, Petah Tikva, Petah Tikva, Israel